CLINICAL TRIAL: NCT06407284
Title: Brighter Bites & Legacy Community Health Produce Rx: Evaluating the Feasibility and Effectiveness of a School-based Clinical Nutrition Program With Produce Prescription
Brief Title: Brighter Bites/Legacy Produce Rx Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: USDA The Gus Schumacher Nutrition Incentive Program (GusNIP) (Unknown)
Responsible Party: Principal Investigator, Ru-Jye Chuang, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-23-0850
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Child Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Produce Prescription Group (Experimental)
  Interventions: Other: Produce Prescription Group
- Control Group (Active Comparator)
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Produce Prescription Group — Participants will receive 16 produce bags, each containing approximately 50 servings of F&V. The produce bags will be assembled by Brighter Bites at school sites using donated produce and delivered to houses using DoorDash. F&V bags will be distributed to families every 2 weeks for 16 distributions (over approximately 32 weeks). Participants will also receive nutrition education, including MyPlate.gov's Start Simple App for adolescents, and a Virtual Culinary Medicine Program for parents; these nutrition education programs are theory-driven, tailored to diverse populations, and proven to support behavior change.
  Arms: Produce Prescription Group
Other: Control Group — Participants in this group will be selected from de-identified Electronic Health Record (EHR) provided by Legacy Community Health with a 1-to-1 match to the intervention group participant's demographic characteristics and Medicaid eligibility.
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess the effectiveness of the produce prescription program at improving weight status and obesity-related health outcomes of participants, to examine the impacts of the program on household food insecurity and nutrition security, to examine the impacts of the program on participating adolescents' dietary behavioral outcomes, their home nutrition environment and feeding practices and to examine the impacts of the program in reducing healthcare use and associated costs

ELIGIBILITY:
Inclusion Criteria:

* Must be a patient at one of the four Legacy Community Health School-based clinics in Galena Park, Texas
* BMI greater than or equal to 85th percentile
* reside within a 10-mile radius of Houston Food Bank
* Medicaid recipients or low-income uninsured
* parents must be able to read and write in English or Spanish to complete surveys
* patient and parents must confirm their willingness to complete the participant's well-child visit for the entire period of the study (approximately one year).

Exclusion Criteria:

* currently participating in Brighter Bites
* with a family member/sibling currently participating in Brighter Bites

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in body mass index (BMI) | baseline , post intervention (32 weeks after baseline)
  This will be collected from chart reviews as these measures are routinely collected for all pediatric patients in this weight classification based on the American Association of Pediatric recommendations.
Change in systolic blood pressure | baseline , post intervention (32 weeks after baseline)
  This will be collected from chart reviews as these measures are routinely collected for all pediatric patients in this weight classification based on the American Association of Pediatric recommendations.
Change in diastolic blood pressure | baseline , post intervention (32 weeks after baseline)
  This will be collected from chart reviews as these measures are routinely collected for all pediatric patients in this weight classification based on the American Association of Pediatric recommendations.
Change in hemoglobin A1c as assessed by blood work | baseline , post intervention (32 weeks after baseline)
  This will be collected from chart reviews as these measures are routinely collected for all pediatric patients in this weight classification based on the American Association of Pediatric recommendations.
Change in Aspartate transaminase (AST) assessed by blood work | baseline , post intervention (32 weeks after baseline)
  This will be collected from chart reviews as these measures are routinely collected for all pediatric patients in this weight classification based on the American Association of Pediatric recommendations.
Change in Alanine transaminase (ALT) assessed by blood work | baseline , post intervention (32 weeks after baseline)
  This will be collected from chart reviews as these measures are routinely collected for all pediatric patients in this weight classification based on the American Association of Pediatric recommendations.
Change in lipid panels assessed by blood work | baseline , post intervention (32 weeks after baseline)
  This will be collected from chart reviews as these measures are routinely collected for all pediatric patients in this weight classification based on the American Association of Pediatric recommendations.

SECONDARY OUTCOMES:
Change in household food insecurity prevalence among participants (measured as a percentage) as assessed by the two item Hunger Vital Sign screening tool | baseline , post intervention (32 weeks after baseline)
  This is a 2 item questionnaire and each is categorically scored as often true, sometimes true or never true, higher number indicating higher prevalence of household food insecurity
Change in household food insecurity as assessed by the U.S. Household Food Security Survey Module: Six-Item Short Form Economic Research Service | baseline , post intervention (32 weeks after baseline)
  This is a 6 item questionnaire and raw scores range from 0-6, higher score indicating worse outcome
Change in nutrition security as assessed by the self reported Perceived Limited Ability validated screener | baseline , post intervention (32 weeks after baseline)
  This is a 4 item questionnaire, each is scored from 0-4, higher score indicating better outcome
Change in amount of fruit and vegetable intake | baseline , post intervention (32 weeks after baseline)
Change in amount of junk food consumed | baseline , post intervention (32 weeks after baseline)
Change in number of times subject eats out at restaurants | baseline , post intervention (32 weeks after baseline)
Change in parent feeding practices as assessed by the number of times parent has cooked food from scratch | baseline , post intervention (32 weeks after baseline)
Change in parent feeding practices as assessed by the number of times parent has used nutrition facts labels to make purchasing decisions | baseline , post intervention (32 weeks after baseline)
Change in parent feeding practices as assessed by the number of times parent has eaten meals with their referent child | baseline , post intervention (32 weeks after baseline)
Change in impact of the Produce Prescription intervention on adolescent patients' behavioral and emotional health as assessed by the Patient Health Questionnaire for Adolescents (PHQ-A) | baseline , post intervention (32 weeks after baseline)
  This is a 9 item questionnaire and each is scored from 0(not at all) to 3(nearly every day), for a maximum score of 27, higher score indicating worse outcome
Healthcare usage as assessed by the number of well-visits | post intervention (32 weeks after baseline)
Healthcare usage as assessed by the number of visits due to illness | post intervention (32 weeks after baseline)
Healthcare usage as assessed by the number of no shows to clinic appointments | From 6 months prior to the intervention to two months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Jye Chuang, DrPH, M.S., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No